CLINICAL TRIAL: NCT03736369
Title: A Multi-Center, Randomized, Double-Blind, Active-controlled, Parallel-Group, Phase 3, Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Erosive Gastroesophageal Reflux Disease (Phase 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP14012301
Record Dates: First submitted 2018-10-26; First posted 2018-11-09 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — fexuprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP14012 40mg (Experimental): Orally, once daily
  Interventions: Drug: DWP14012 40mg; Drug: Esomeprazole 40mg placebo
- Esomeprazole 40mg (Active Comparator): Orally, once daily
  Interventions: Drug: DWP14012 40mg placebo; Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: DWP14012 40mg — DWP14012 40mg, tablet, orally, once daily for up to 8 weeks
  Arms: DWP14012 40mg
Drug: DWP14012 40mg placebo — DWP14012 40mg placebo-matching tablet, orally, once daily for up to 8 weeks
  Arms: Esomeprazole 40mg
Drug: Esomeprazole 40mg — Esomeprazole 40mg tablet, orally, once daily for up to 8 weeks
  Other Names: Nexium 40mg
  Arms: Esomeprazole 40mg
Drug: Esomeprazole 40mg placebo — Esomeprazole 40mg placebo-matching tablet, orally, once daily for up to 8 weeks
  Other Names: Nexium 40mg placebo
  Arms: DWP14012 40mg

SUMMARY:
The purpose of study is to confirm the efficacy of DWP14012 Xmg, Once daily, compared to esomeprazole 40mg in patients with erosive gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 and 75 years old based on the date of written agreement
* Those who have been diagnosed with erosive gastroesophageal reflux disease(EGRD) of LA Grade A-D on the upper gastrointestinal endoscopy
* Those who experienced symptoms of heartburn or acid regurgitation within the last 7 days

Exclusion Criteria:

* Those who have undergone gastric acid suppression or gastric, esophageal surgery
* Those who with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Cumulative healing rate of erosive esophagitis at 8week by endoscopy | at 8week

SECONDARY OUTCOMES:
Cumulative healing rate of erosive esophagitis at 4week by endoscopy | at 4week
Reflux disease symptom assessment using RDQ(Reflux disease questionnaire) | at 4week and 8week
  Mean change of the frequency or severity of main symptoms
Quality of Life assessment using GERD-HRQL(GERD-Health related quality life) | at 4week and 8week
  Mean change of the total score of GERD-HRQL

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No